CLINICAL TRIAL: NCT05604092
Title: White Matter Lesion Load and Location in Relation to Cognition, Fatigue and Physical Disability in Patients With Relapsing Remitting Multiple Sclerosis
Brief Title: Lesion Load and Location in Relation to Cognition, Fatigue and Physical Disability in RRMS
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, professor, Assiut University
Other Study IDs: lesion load and distribution
Record Dates: First submitted 2022-10-21; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: VolBrain, a fully automated platform to generate the volumetric data (lesion count, volume and location as well as different atrophy measures) — VolBrain, a fully automated platform that uses anonymized compressed NIFTI files to generate the volumetric data. Volbrain is increasingly recognized and compared to other volumetric tools. LesionBrain is a pipeline to automatically segment WM-L from T1 and FLAIR data. Number of lesions, absolute total lesion volume (in cubic cm), normalized lesion volume (percentage of total lesion volume to whole brain volume), lesion burden (percentage of total WM lesion volume to WM volume), and location (Periventricular, Juxtacortical, and Infratentorial) were obtained.
Other: Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) — It includes the Symbol Digit Modalities Test (SDMT) for evaluating the information processing speed, the California Verbal Learning Test (CVLT-II) for evaluating verbal learning and memory, and the Brief Visual Memory Test (BVMT) for evaluating visual learning and memory. Cut off values were calculated as 1.5 SD below mean according to a group of healthy individuals who are matched in age, sex and education as following: 22 for SDMT, 38 for CVLT, and 10 for BVMTR

SUMMARY:
In relapsing remitting multiple sclerosis (RRMS) the relationship between cognitive impairment (CI), fatigue and physical disability with white matter lesion load (WM-LL), location among other volumetric measures using automated platforms is still unclear.

DETAILED DESCRIPTION:
Cognitive impairment (CI) and fatigue have been recognized as an important feature of MS, affecting up to 70% patients (1), evident since onset and increase in both prevalence and severity as the disease progresses (2). In fact, their effects on patients and even their caregivers are more pronounced than clinical disability, causing unemployment, treatment non-adherence, personality changes as well as several psychosocial dysfunctions (3-5). Therefore, beside evaluating the physical disability, it is essential for health professionals to objectively evaluate either the cognitive function or fatigue at both baseline and during routine follow up visits for early detection and management (6). Through the advances in MRI techniques and availability of a number of automated software, quantitative radiological assessments became more readily available and feasible in daily practice (7) allowing objective longitudinal monitoring of patients (8,9). Although burden and location of lesions in RRMS is thought to be associated with cognitive impairment (CI), fatigue and physical disability, some controversy results were obtained from previous studies. So, by conducting this study, we aimed at exploring the relationship between different parameters of lesion load and location with fatigue, cognitive and physical disability in RRMS patients.

ELIGIBILITY:
Inclusion Criteria:

* : adult patients of both sexes diagnosed with RRMS according to 2017 McDonald diagnostic criteria

Exclusion Criteria:

* Patients with relapse or steroid administration in the past 30 days were excluded. Patients who have any medical conditions that may affect cognition, and those on psychoactive pharmacotherapy were also excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with relapsing remitting multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
The relation of white matter lesion load, location and parameters of cognitive function measured by BICAMS | 6 months
  correlation of BICAMS subtests scores to different parameters of white matter lesion load, distribution and load (volume and number of lesion) measurements (whole brain atrophy, grey matter and white matter lesion load) to identify best predictors of cognitive impairment
The relation of white matter lesion load, location and Fatigue in patients with relapsing remitting multiple sclerosis | 6 months
  correlation between fatigue severity, with white matter lesion load, and distribution in order to identify predictors of fatigue

SECONDARY OUTCOMES:
the relation of white matter lesion load, location and atrophy parameters to physical disability in patients with relapsing remitting multiple sclerosis | 6 months
  correlation of EDSS scores, with white matter lesion load and distribution

CONTACTS AND LOCATIONS:
Overall Officials: Eman M Khedr, professor, Principal Investigator — Assuit university hospital
Locations (1):
- Eman Khedr, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No